CLINICAL TRIAL: NCT00816725
Title: Using the Internet for English/Spanish Randomized Trials for Postpartum Depression
Brief Title: Effectiveness of a Web-based Prevention Program for Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alinne Barrera, Staff Psychologist, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F32MH077371 (NIH); F32MH077371 (NIH); 5A; DATR AK-TAIF (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Depression; Postpartum Depression
Keywords: Postnatal Depression; Cognitive Behavioral Therapy; Mood Management; Self-help; Internet
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-help course and information (Experimental)
  Interventions: Behavioral: Mothers and babies Internet course and PPD informational brochure

INTERVENTIONS:
Behavioral: Mothers and babies Internet course and PPD informational brochure — An eight-lesson, self-help, Web-based program for the prevention of postpartum depression based on cognitive behavioral therapy, social-learning, and attachment theory. The PPD informational brochure is a four-page pamphlet that contains information about postpartum depression.

SUMMARY:
The original trial will evaluate the effectiveness of a Web-based program in preventing postpartum depression. The site has been modified to provide materials from both conditions.

DETAILED DESCRIPTION:
Depression is a mental health condition in which symptoms such as sadness, inability to feel pleasure, and loss of energy interfere with a person's normal life. Postpartum depression is a type of depression experienced by women after giving birth to a child. In this study an intervention for preventing postpartum depression that has been adapted for use over the Internet will be tested. Administering a depression-prevention program over the Internet has several advantages: after the initial investment is made to develop the program, costs are lower for treating each patient; online treatment is more accessible to a greater number of people than any given clinic; and participants who may be worried about a stigma associated with mental health problems often feel more comfortable seeking information through the Internet. Previous research has shown that symptoms of depression can be reduced through Internet-based interventions, but no research has examined such interventions specifically for postpartum depression. The program tested in this study is not aimed at replacing in-person mental health care-in fact, people who have signs of serious depression will be directed to in-person mental health care. Instead, the program is aimed at providing an additional mental health service among the range of available options.

The original trial was a two-arm pilot prevention of postpartum depression trial comparing the Internet-based course called "Mothers and Babies/Mamás y Bebés" (M&B) to informational materials on postpartum depression. In the original trial, 1088 pregnant women were recruited and randomized (as anticipated) to either condition. The study Website has therefore been modified such that all participants who consent to participate will now receive materials from both conditions. We have eliminated the randomization procedure.

As in the original study, participants be allowed to enroll at any time during their pregnancies and will be followed for 6 months after the birth of their children, so the length of participation will vary between 6 and 15 months. After undergoing a screening process, participants will now have access to both the Internet-based course called "Mothers and Babies/Mamás y Bebés" (M&B) and the informational materials. The informational materials will include information about postpartum depression and depression that may occur before childbirth. All participants will be invited via email to complete monthly assessments for the duration of the study. These assessments will measure mood, depression, and satisfaction with the assigned intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Fluent in English or Spanish

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Measured monthly for 6 months postpartum

SECONDARY OUTCOMES:
Center for Epidemiologic Studies-Depression (CES-D) Scale | Measured monthly for 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Alinne Z. Barrera, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Barrera AZ, Kelman AR, Munoz RF. Keywords to recruit Spanish- and English-speaking participants: evidence from an online postpartum depression randomized controlled trial. J Med Internet Res. 2014 Jan 9;16(1):e6. doi: 10.2196/jmir.2999. PMID 24407163